CLINICAL TRIAL: NCT00972816
Title: A Pivotal Randomized, Single-Blind, Dose-Finding Study to Evaluate Immunogenicity, Safety and Tolerability of Different Formulations of an Adjuvanted and Non-Adjuvanted Egg-Derived, Inactivated Novel Swine Origin A/H1N1 Monovalent Subunit Influenza Virus Vaccine in Healthy Pediatric Subjects 3 to < 9 Years of Age
Brief Title: Safety and Immunogenicity of A/H1N1-SOIV (Swine Flu) Vaccine With and Without Adjuvant in Children (3 to < 9 Years)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: V112_02
Record Dates: First submitted 2009-09-02; First posted 2009-09-09 (Estimated); Results first posted 2011-01-27 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-03

CONDITIONS: Influenza
Keywords: Swine Flu; Flu; Vaccine; Children; Adjuvant
MeSH Terms: conditions — Influenza, Human; Orthomyxoviridae Infections

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (8):
- 3.75_(50)MF59 (Experimental): 3.75 μg A/H1N1 antigen with 50% MF59 adjuvant administered on study day 1 and day 22
  Interventions: Biological: MF59-eH1N1
- 7.5_(0) MF59 (Experimental): 7.5 μg A/H1N1 antigen without MF59 adjuvant administered on study day 1 and day 22
  Interventions: Biological: MF59-eH1N1
- 7.5_(50) MF59 (Experimental): 7.5 μg A/H1N1 antigen with 50% MF59 adjuvant administered on study day 1 and day 22
  Interventions: Biological: MF59-eH1N1
- 7.5_(100) MF59 (Experimental): 7.5 μg A/H1N1 antigen with 100% MF59 adjuvant administered on study day 1 and day 22
  Interventions: Biological: MF59-eH1N1
- 15_(0) MF59 (Experimental): 15 μg A/H1N1 antigen without MF59 adjuvant administered on study day 1 and day 22
  Interventions: Biological: MF59-eH1N1
- 15_(50)MF59 (Experimental): 15 μg A/H1N1 antigen with 50% MF59 adjuvant administered on study day 1 and day 22
  Interventions: Biological: MF59-eH1N1
- 15_(100) MF59 (Experimental): 15 μg A/H1N1 antigen with 100% MF59 adjuvant administered on study day 1 and day 22
  Interventions: Biological: MF59-eH1N1
- 30_(0) MF59 (Experimental): 30 μg A/H1N1 antigen without MF59 adjuvant administered on study day 1 and day 22
  Interventions: Biological: MF59-eH1N1

INTERVENTIONS:
Biological: MF59-eH1N1 — MF59 adjuvanted with egg-derived A/H1N1 antigen. MF59-eH1N1 vaccine is the same vaccine as A/H1N1-SOIV (Swine Origin A/H1N1 Influenza Virus).

SUMMARY:
This study will evaluate the safety and immunogenicity of different combinations of A/H1N1 S-OIV (swine flu) vaccine in healthy young children.

ELIGIBILITY:
Inclusion Criteria:

* Children 3 to < 9 years of age in good health as determined by medical history, physical assessment and clinical judgement of the investigator and without influenza within the past 6 months.

Exclusion Criteria:

* History of serious disease.
* History of serious reaction following administration of vaccine or hypersensitivity to vaccine components.
* Known or suspected impairment/alteration of immune function.
* Receipt or planned receipt of seasonal trivalent influenza vaccine within 1 week before or after each study vaccination.

For additional entry criteria, please refer to protocol.

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1357 (Actual)
Dates: Start 2009-09; Primary Completion 2009-11 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines and Diagnostics, Study Director — Novartis
Locations (35):
- United States (34):
  - Premier Health Research Center, LLC, Downey, California
  - Madera Family Medical Group, Madera, California
  - Center for Clincal Trials, LLC, Paramount, California
  - Center for Clinical Trials, LLC, Paramount, California
  - Center for Clinical Trials of San Gabriel, West Covina, California
  - 1st International Research Centers, Thornton, Colorado
  - Pediatrics and Adolescent Medicine, Marietta, Georgia
  - Pediatrics and Adolescent Medicine, Woodstock, Georgia
  - Northern Illinois Research Associates, DeKalb, Illinois
  - Bluegrass Clinical Research, Inc., New Albany, Indiana
  - Heartland Research Associates LLC, Arkansas City, Kansas
  - Heartland Research Associates LLC, Newton, Kansas
  - Bluegrass Clinical Research, Inc (Brownsboro for drug shipment), Louisville, Kentucky
  - Meridien Clinical Research, Omaha, Nebraska
  - Clinical Research Center of Nevada, Henderson, Nevada
  - Capital Pediatrics and Adolescent Ctr., Raleigh, North Carolina
  - Dr. Senders and Associates, Pediatrics, Cleveland, Ohio
  - Prestige Clinical Research, Franklin, Ohio
  - IPS Research, Oklahoma City, Oklahoma
  - The Portland Clinic LLP, Beaverton, Oregon
  - Children's Health Care -West, Erie, Pennsylvania
  - UPMC/Community Medicine (pediatrics), Greenville, Pennsylvania
  - Pediatric Physicians Research, Inc., Jefferson Hills, Pennsylvania
  - Pediatric Alliance - Greentree Division (pediatrics), Pittsburgh, Pennsylvania
  - Omega Clinical Research, Warwick, Rhode Island
  - Holston Medical Group, Kingsport, Tennessee
  - Research Across America, Dallas, Texas
  - West Houston Clinical Research Service, Houston, Texas
  - Pediatric Healthcare of NW Houston, Tomball, Texas
  - J.Lewis Research, Inc./Foothill Family Clinic, Salt Lake City, Utah
  - J. Lewis Research, Inc./Foothill Family Clinic South, Salt Lake City, Utah
  - PI-Coor Clinical Research, Burke, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - Rockwood Research Center, Spokane, Washington
- Instituto Nacional de Ciencias, Tlalpan, Mexico City, Mexico

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 36 centers in the U.S., of which 34 centers enrolled subjects.
Groups:
- 3.75_(50) MF59: 3.75 μg A/H1N1 antigen with 50% MF59 adjuvant administered on study day 1 and day 22
- 7.5_(50)MF59: 7.5 μg A/H1N1 antigen with 50% MF59 adjuvant administered on study day 1 and day 22
- 7.5_(100)MF59: 7.5 μg A/H1N1 antigen with 100% MF59 adjuvant administered on study day 1 and day 22
- 15_(50) MF59: 15 μg A/H1N1 antigen with 50% MF59 adjuvant administered on study day 1 and day 22
Period: Overall Study
Arm/Group | 3.75_(50) MF59 | 7.5_(0) MF59 | 7.5_(50)MF59 | 7.5_(100)MF59 | 15_(0) MF59 | 15_(50) MF59 | 15_(100) MF59 | 30_(0) MF59
Started | 173 | 169 | 169 | 169 | 169 | 169 | 169 | 170
Completed | 156 | 158 | 160 | 161 | 157 | 158 | 159 | 161
Not Completed | 17 | 11 | 9 | 8 | 12 | 11 | 10 | 9
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 2 | 1 | 3 | 0 | 1 | 1 | 2
Not completed — Lost to Follow-up | 11 | 9 | 7 | 5 | 11 | 10 | 7 | 7
Not completed — Inappropriate enrolment | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Not completed — Unable to classify | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- 3.75_(50)MF59: 50% of MF59 with 3.75 µg A/H1N1 antigen
- 7.5 Without MF59: 1 dose of 7.5 µg A/H1N1
- 7.5_(50)MF59: 50% of MF59 with 7.5 µg A/H1N1 antigen
- 7.5_(100)MF59: 100% of MF59 with 7.5 µg A/H1N1 antigen
- 15 Without MF59: 1 dose of 15 µg A/H1N1
- 15_(50)MF59: 50% of MF59 with 15 µg A/H1N1 antigen
- 15_(100)MF59: 100% of MF59 with 15 µg A/H1N1 antigen
- 30 Without MF59: 1 dose of 30 µg A/H1N1
- Total: Total of all reporting groups
Arm/Group | 3.75_(50)MF59 | 7.5 Without MF59 | 7.5_(50)MF59 | 7.5_(100)MF59 | 15 Without MF59 | 15_(50)MF59 | 15_(100)MF59 | 30 Without MF59 | Total
Number analyzed (Participants) | 173 | 169 | 169 | 169 | 169 | 169 | 169 | 170 | 1357
Age, Continuous [Mean (Standard Deviation); unit: years] | 5.6 (1.7) | 5.2 (1.7) | 5.5 (1.8) | 5.9 (1.7) | 5.6 (1.7) | 5.5 (1.7) | 5.5 (1.7) | 5.5 (1.7) | 5.5 (1.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81 | 88 | 83 | 83 | 79 | 80 | 75 | 83 | 652
  Male | 92 | 81 | 86 | 86 | 90 | 89 | 94 | 87 | 705

OUTCOME MEASURES:

1. Primary Outcome: Antibody Responses According to the Hemagglutinin Inhibition (HI) Assay After the First and Second Vaccinations
Description: HI antibody assay (used to assess immune responses in subjects following vaccination) according to the Center for Biologics Evaluation and Research (CBER) guidance for <65 years of age: The lower bound of the two-sided 95% Confidence Interval (CI) for the percentages of subjects achieving seroconversion for HI antibody should be ≥ 40% and the lower bound of the two-sided 95% CI for the percentages of subjects achieving an HI antibody titer ≥ 1:40 should be ≥ 70%. Both criteria (seroconversion and HI antibody titer ≥ 40) had to be fulfilled to establish immunogenicity.
  PPS Day 1-29 analysis set: N= 143, 149, 149, 146, 147, 147, 144, and 144 for Groups A, B, C, D, E, F,G,and H respectively.
  PPS Day 1-202 analysis set: N= 82, 85, 84, 84, 86, 87, 82, and 79 for Groups A, B, C, D, E, F, G, and H respectively.
  PPS Day 1-387 analysis set: N= 55, 63, 61, 58, 61, 65, 59, and 63 for Groups A, B, C, D, E, F, G, and H respectively.
Time Frame: Day 22, Day 29, Day 43, Day 202 and Day 387
Population: The analysis was performed on per protocol set (PPS) population
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | 3.75_(50)MF59 | 7.5 Without MF59 | 7.5_(50)MF59 | 7.5_(100)MF59 | 15 Without MF59 | 15_(50)MF59 | 15_(100)MF59 | 30 Without MF59
Number analyzed (Participants) | 152 | 156 | 156 | 156 | 155 | 157 | 156 | 153
percentage of subjects
  HI titer ≥1:40 (Baseline) | 11 [6 to 17] | 9 [5 to 15] | 13 [8 to 19] | 11 [6 to 170] | 15 [10 to 22] | 9 [5 to 15] | 8 [4 to 13] | 12 [8 to 19]
  HI titer ≥1:40 day 22 | 84 [77 to 89] | 48 [40 to 56] | 81 [74 to 87] | 91 [85 to 95] | 61 [52 to 68] | 82 [75 to 88] | 94 [89 to 97] | 65 [57 to 73]
  Seroconversion day 22 | 82 [74 to 87] | 46 [38 to 54] | 78 [70 to 84] | 88 [82 to 93] | 58 [50 to 66] | 82 [75 to 87] | 92 [86 to 95] | 60 [52 to 68]
  HI titer ≥1:40 (Day 29) | 99 [96 to 100] | 79 [71 to 85] | 100 [98 to 100] | 99 [95 to 100] | 88 [82 to 93] | 100 [98 to 100] | 100 [97 to 100] | 97 [92 to 99]
  Seroconversion (Day 29) | 99 [95 to 100] | 78 [70 to 84] | 99 [95 to 100] | 99 [95 to 100] | 87 [81 to 92] | 100 [98 to 100] | 100 [97 to 100] | 94 [88 to 97]
  HI titer ≥1:40 day 43 | 99 [96 to 100] | 79 [72 to 85] | 100 [98 to 100] | 99 [95 to 100] | 87 [81 to 92] | 99 [97 to 100] | 100 [98 to 100] | 92 [86 to 95]
  Seroconversion day 43 | 98 [94 to 100] | 78 [70 to 84] | 97 [93 to 99] | 97 [94 to 99] | 85 [78 to 90] | 99 [95 to 100] | 99 [96 to 100] | 88 [82 to 93]
  HI titer ≥1:40 day 202 (N=82,85,84,84,86,87,82,79) | 95 [88 to 99] | 65 [54 to 75] | 93 [85 to 97] | 95 [88 to 99] | 74 [64 to 83] | 95 [89 to 99] | 95 [88 to 99] | 81 [71 to 89]
  Seroconversion day 202 (N=82,85,84,84,86,87,82,79) | 83 [73 to 90] | 55 [44 to 66] | 83 [74 to 91] | 83 [74 to 91] | 63 [52 to 73] | 90 [81 to 95] | 90 [82 to 96] | 66 [54 to 76]
  HI titer ≥1:40 day 387 (N=55,63,61,58,61,65,59,63) | 80 [67 to 90] | 56 [42 to 68] | 75 [63 to 86] | 88 [77 to 95] | 49 [36 to 62] | 78 [67 to 88] | 81 [69 to 90] | 65 [52 to 77]
  Seroconversion day 387 (N=55,63,61,58,61,65,59,63) | 65 [51 to 78] | 49 [36 to 62] | 69 [56 to 80] | 78 [65 to 87] | 44 [32 to 58] | 75 [63 to 85] | 71 [58 to 82] | 51 [38 to 64]

2. Secondary Outcome: Geometric Mean Titer (GMT) After Each Vaccination by Vaccine Group
Description: Immunogenicity was measured in terms of GMTs After each vaccination by vaccine Group.
  PPS Day1-29 analysis set: N=143, 149, 149, 146, 147, 147, 144, and 144 for Groups A, B, C, D, E, F, G, and H respectively.
  PPS Day 1-202 analysis set. N= 82, 85, 84, 84, 86, 87, 82, and 79 for Groups A, B, C, D, E, F, G, and H respectively.
Time Frame: Day 22, Day 29, Day 43, Day 202 and Day 387
Population: The analysis was performed on per protocol set (PPS) population
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | 3.75_(50)MF59 | 7.5 Without MF59 | 7.5_(50)MF59 | 7.5_(100)MF59 | 15 Without MF59 | 15_(50)MF59 | 15_(100)MF59 | 30 Without MF59
Number analyzed (Participants) | 152 | 156 | 156 | 156 | 155 | 157 | 156 | 153
Titers
  GMT Baseline | 8.5 [7 to 10] | 7.3 [6 to 8.8] | 8.7 [7.2 to 11] | 8.7 [6.7 to 9.9] | 9.1 [7.5 to 11] | 7.5 [6.2 to 9.1] | 7 [5.8 to 8.4] | 9.1 [7.5 to 11]
  GMTs day 22 | 107 [78 to 148] | 27 [20 to 37] | 88 [64 to 121] | 163 [118 to 223] | 49 [36 to 68] | 106 [77 to 145] | 160 [116 to 220] | 62 [45 to 85]
  GMT Day 29 | 747 [588 to 950] | 138 [109 to 174] | 685 [542 to 866] | 984 [775 to 1249] | 214 [169 to 271] | 761 [600 to 966] | 1070 [841 to 1360] | 297 [235 to 377]
  GMTs day 43 | 560 [450 to 699] | 113 [91 to 140] | 480 [386 to 597] | 637 [511 to 793] | 174 [140 to 217] | 524 [420 to 652] | 778 [625 to 969] | 223 [179 to 278]
  GMTs day 202 (N=143,149,149,146,147,147,144,144) | 117 [88 to 157] | 45 [34 to 59] | 107 [80 to 144] | 132 [99 to 177] | 55 [41 to 74] | 134 [100 to 179] | 131 [97 to 176] | 81 [60 to 109]
  GMTs day 387 (N=55,63,61,58,61,65,59,63) | 54 [37 to 78] | 28 [20 to 40] | 57 [40 to 82] | 70 [49 to 102] | 30 [21 to 42] | 59 [41 to 83] | 63 [44 to 90] | 45 [31 to 64]
Statistical Analysis 1: Comparison: 3.75_(50)MF59 vs 7.5 Without MF59; A difference was assumed to be statistically significant if the 2-sided 95% CI around the ratio of GMTs did not contain 1, in which case one group is either statistically significantly superior or statistically inferior to the other; Test type: Non-Inferiority or Equivalence — For pairwise vaccine group compared, least squares GMT and associated 2-sided 95% CI, median, minimum, and maximum HI titer values were determined. The two-sided 95% CIs was calculated and assessed against a non-inferiority margin of 0.5. Subsequently the same non-inferiority hypothesis was tested using a non-inferiority margin of 0.67; Geometric mean ratio at day 22 = 3.998, 95% CI 2-sided [2.659 to 6.009]
Statistical Analysis 2: Comparison: 3.75_(50)MF59 vs 7.5_(50)MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio at day 22 = 1.222, 95% CI 2-sided [0.813 to 1.838]
Statistical Analysis 3: Comparison: 3.75_(50)MF59 vs 7.5_(100)MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio at day 22 = 0.661, 95% CI 2-sided [0.440 to 0.994]
Statistical Analysis 4: Comparison: 3.75_(50)MF59 vs 15 Without MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio at day 22 = 2.178, 95% CI 2-sided [1.449 to 3.276]
Statistical Analysis 5: Comparison: 3.75_(50)MF59 vs 15_(50)MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio at day 22 = 1.017, 95% CI 2-sided [0.676 to 1.528]
Statistical Analysis 6: Comparison: 3.75_(50)MF59 vs 15_(100)MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio at day 22 = 0.673, 95% CI 2-sided [0.448 to 1.012]
Statistical Analysis 7: Comparison: 3.75_(50)MF59 vs 30 Without MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio at day 22 = 1.742, 95% CI 2-sided [1.156 to 2.626]
Statistical Analysis 8: Comparison: 7.5 Without MF59 vs 7.5_(50)MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio at day 22 = 0.306, 95% CI 2-sided [0.204 to 0.458]
Statistical Analysis 9: Comparison: 7.5 Without MF59 vs 7.5_(100)MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio at day 22 = 0.165, 95% CI 2-sided [0.110 to 0.248]
Statistical Analysis 10: Comparison: 7.5 Without MF59 vs 15 Without MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio at day 22 = 0.545, 95% CI 2-sided [0.363 to 0.818]
Statistical Analysis 11: Comparison: 7.5 Without MF59 vs 15_(50)MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio at day 22 = 0.254, 95% CI 2-sided [0.170 to 0.381]
Statistical Analysis 12: Comparison: 7.5 Without MF59 vs 15_(100)MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio at day 22 = 0.168, 95% CI 2-sided [0.112 to 0.252]
Statistical Analysis 13: Comparison: 7.5 Without MF59 vs 30 Without MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio at day 22 = 0.436, 95% CI 2-sided [0.290 to 0.655]
Statistical Analysis 14: Comparison: 7.5_(50)MF59 vs 7.5_(100)MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio at day 22 = 0.541, 95% CI 2-sided [0.361 to 0.811]
Statistical Analysis 15: Comparison: 7.5_(50)MF59 vs 15 Without MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio at day 22 = 1.783, 95% CI 2-sided [1.188 to 2.676]
Statistical Analysis 16: Comparison: 7.5_(50)MF59 vs 15_(50)MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio at day 22 = 0.832, 95% CI 2-sided [0.555 to 1.246]
Statistical Analysis 17: Comparison: 7.5_(50)MF59 vs 15_(100)MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio at day 22 = 0.551, 95% CI 2-sided [0.367 to 0.826]
Statistical Analysis 18: Comparison: 7.5_(50)MF59 vs 30 Without MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio at day 22 = 1.426, 95% CI 2-sided [0.950 to 2.140]
Statistical Analysis 19: Comparison: 7.5_(100)MF59 vs 15 Without MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio at day 22 = 3.295, 95% CI 2-sided [2.196 to 4.944]
Statistical Analysis 20: Comparison: 7.5_(100)MF59 vs 15_(50)MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio at day 22 = 1.538, 95% CI 2-sided [1.026 to 2.303]
Statistical Analysis 21: Comparison: 7.5_(100)MF59 vs 15_(100)MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio at day 22 = 1.018, 95% CI 2-sided [0.679 to 1.526]
Statistical Analysis 22: Comparison: 7.5_(100)MF59 vs 30 Without MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio at day 22 = 2.635, 95% CI 2-sided [1.754 to 3.959]
Statistical Analysis 23: Comparison: 15 Without MF59 vs 15_(50)MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio at day 22 = 0.467, 95% CI 2-sided [0.311 to 0.7]
Statistical Analysis 24: Comparison: 15 Without MF59 vs 15_(100)MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio at day 22 = 0.309, 95% CI 2-sided [0.206 to 0.463]
Statistical Analysis 25: Comparison: 15 Without MF59 vs 30 Without MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio at day 22 = 0.8, 95% CI 2-sided [0.532 to 1.203]
Statistical Analysis 26: Comparison: 15_(50)MF59 vs 15_(100)MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio at day 22 = 0.662, 95% CI 2-sided [0.442 to 0.992]
Statistical Analysis 27: Comparison: 15_(50)MF59 vs 30 Without MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio at day 22 = 1.714, 95% CI 2-sided [1.142 to 2.572]
Statistical Analysis 28: Comparison: 15_(100)MF59 vs 30 Without MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — A difference was assumed to be statistically significant if the 2-sided 95% CI around the ratio of GMTs did not contain 1, in which case one group is either statistically significantly superior or statistically inferior to the other; Geometric mean ratio at day 22 = 2.589, 95% CI 2-sided [1.723 to 3.889]
Statistical Analysis 29: Comparison: 3.75_(50)MF59 vs 7.5 Without MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio at day 43 = 4.975, 95% CI 2-sided [3.757 to 6.589]
Statistical Analysis 30: Comparison: 3.75_(50)MF59 vs 7.5_(50)MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio at day 43 = 1.168, 95% CI 2-sided [0.881 to 1.547]
Statistical Analysis 31: Comparison: 3.75_(50)MF59 vs 7.5_(100)MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio at day 43 = 0.880, 95% CI 2-sided [0.665 to 1.166]
Statistical Analysis 32: Comparison: 3.75_(50)MF59 vs 15 Without MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio at day 43 = 3.219, 95% CI 2-sided [2.430 to 4.264]
Statistical Analysis 33: Comparison: 3.75_(50)MF59 vs 15_(50)MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio at day 43 = 1.070, 95% CI 2-sided [0.808 to 1.417]
Statistical Analysis 34: Comparison: 3.75_(50)MF59 vs 15_(100)MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio at day 43 = 0.720, 95% CI 2-sided [0.544 to 0.954]
Statistical Analysis 35: Comparison: 3.75_(50)MF59 vs 30 Without MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio at day 43 = 2.509, 95% CI 2-sided [1.891 to 3.330]
Statistical Analysis 36: Comparison: 7.5 Without MF59 vs 7.5_(50)MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio at day 43 = 0.235, 95% CI 2-sided [0.178 to 0.310]
Statistical Analysis 37: Comparison: 7.5 Without MF59 vs 7.5_(100)MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio at day 43 = 0.177, 95% CI 2-sided [0.134 to 0.234]
Statistical Analysis 38: Comparison: 7.5 Without MF59 vs 15 Without MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio at day 43 = 0.647, 95% CI 2-sided [0.489 to 0.856]
Statistical Analysis 39: Comparison: 7.5 Without MF59 vs 15_(50)MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio at day 43 = 0.215, 95% CI 2-sided [0.163 to 0.284]
Statistical Analysis 40: Comparison: 7.5 Without MF59 vs 15_(100)MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio at day 43 = 0.145, 95% CI [0.109 to 0.191]
Statistical Analysis 41: Comparison: 7.5 Without MF59 vs 30 Without MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio at day 43 = 0.504, 95% CI 2-sided [0.381 to 0.668]
Statistical Analysis 42: Comparison: 7.5_(50)MF59 vs 7.5_(100)MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio at day 43 = 0.754, 95% CI 2-sided [0.570 to 0.997]
Statistical Analysis 43: Comparison: 7.5_(50)MF59 vs 15 Without MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio at day 43 = 2.756, 95% CI 2-sided [2.083 to 3.647]
Statistical Analysis 44: Comparison: 7.5_(50)MF59 vs 15_(50)MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio at day 43 = 0.916, 95% CI 2-sided [0.694 to 1.211]
Statistical Analysis 45: Comparison: 7.5_(50)MF59 vs 15_(100)MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio at day 43 = 0.616, 95% CI 2-sided [0.466 to 1.815]
Statistical Analysis 46: Comparison: 7.5_(50)MF59 vs 30 Without MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio at day 43 = 2.149, 95% CI 2-sided [1.624 to 2.843]
Statistical Analysis 47: Comparison: 7.5_(100)MF59 vs 15 Without MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio at day 43 = 3.656, 95% CI 2-sided [2.764 to 4.836]
Statistical Analysis 48: Comparison: 7.5_(100)MF59 vs 15_(50)MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio at day 43 = 1.216, 95% CI 2-sided [0.920 to 1.606]
Statistical Analysis 49: Comparison: 7.5_(100)MF59 vs 15_(100)MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio at day 43 = 0.818, 95% CI 2-sided [0.619 to 1.081]
Statistical Analysis 50: Comparison: 7.5_(100)MF59 vs 30 Without MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio at day 43 = 2.850, 95% CI 2-sided [2.152 to 3.773]
Statistical Analysis 51: Comparison: 15 Without MF59 vs 15_(50)MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio at day 43 = 0.332, 95% CI 2-sided [0.251 to 0.440]
Statistical Analysis 52: Comparison: 15 Without MF59 vs 15_(100)MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio at day 43 = 0.224, 95% CI 2-sided [0.169 to 0.296]
Statistical Analysis 53: Comparison: 15 Without MF59 vs 30 Without MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio at day 43 = 0.780, 95% CI 2-sided [0.588 to 1.003]
Statistical Analysis 54: Comparison: 15_(50)MF59 vs 15_(100)MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio at day 43 = 0.673, 95% CI 2-sided [0.509 to 0.889]
Statistical Analysis 55: Comparison: 15_(50)MF59 vs 30 Without MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio at day 43 = 2.345, 95% CI 2-sided [1.772 to 3.102]
Statistical Analysis 56: Comparison: 15_(100)MF59 vs 30 Without MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio at day 43 = 3.485, 95% CI 2-sided [2.633 to 4.614]
Statistical Analysis 57: Comparison: 3.75_(50)MF59 vs 7.5 Without MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio at day 202 = 2.624, 95% CI 2-sided [1.817 to 3.789]
Statistical Analysis 58: Comparison: 3.75_(50)MF59 vs 7.5_(50)MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio at day 202 = 1.096, 95% CI 2-sided [0.760 to 1.580]
Statistical Analysis 59: Comparison: 3.75_(50)MF59 vs 7.5_(100)MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio at day 202 = 0.888, 95% CI 2-sided [0.615 to 1.282]
Statistical Analysis 60: Comparison: 3.75_(50)MF59 vs 15 Without MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio at day 202 = 2.120, 95% CI 2-sided [1.473 to 3.052]
Statistical Analysis 61: Comparison: 3.75_(50)MF59 vs 15_(50)MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio at day 202 = 0.876, 95% CI 2-sided [0.610 to 1.260]
Statistical Analysis 62: Comparison: 3.75_(50)MF59 vs 15_(100)MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio at day 202 = 0.898, 95% CI 2-sided [0.622 to 1.298]
Statistical Analysis 63: Comparison: 3.75_(50)MF59 vs 30 Without MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio at day 202 = 1.451, 95% CI 2-sided [1.000 to 2.105]
Statistical Analysis 64: Comparison: 7.5 Without MF59 vs 7.5_(50)MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio at day 202 = 0.418, 95% CI 2-sided [0.289 to 0.603]
Statistical Analysis 65: Comparison: 7.5 Without MF59 vs 7.5_(100)MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio at day 202 = 0.338, 95% CI 2-sided [0.235 to 0.487]
Statistical Analysis 66: Comparison: 7.5 Without MF59 vs 15 Without MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio at day 202 = 0.808, 95% CI 2-sided [0.561 to 1.165]
Statistical Analysis 67: Comparison: 7.5 Without MF59 vs 15 Without MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio at day 202 = 0.334, 95% CI 2-sided [0.233 to 0.479]
Statistical Analysis 68: Comparison: 7.5 Without MF59 vs 15_(100)MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio at day 202 = 0.342, 95% CI 2-sided [0.237 to 0.494]
Statistical Analysis 69: Comparison: 7.5 Without MF59 vs 30 Without MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio at day 202 = 0.553, 95% CI 2-sided [0.382 to 0.801]
Statistical Analysis 70: Comparison: 7.5_(50)MF59 vs 7.5_(100)MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio at day 202 = 0.811, 95% CI 2-sided [0.562 to 1.169]
Statistical Analysis 71: Comparison: 7.5_(50)MF59 vs 15 Without MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio at day 202 = 1.935, 95% CI 2-sided [1.347 to 2.780]
Statistical Analysis 72: Comparison: 7.5_(50)MF59 vs 15_(50)MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio at day 202 = 0.800, 95% CI 2-sided [0.558 to 1.147]
Statistical Analysis 73: Comparison: 7.5_(50)MF59 vs 15_(100)MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio at day 202 = 0.820, 95% CI 2-sided [0.568 to 1.184]
Statistical Analysis 74: Comparison: 7.5_(50)MF59 vs 30 Without MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio at day 202 = 1.324, 95% CI 2-sided [0.915 to 1.917]
Statistical Analysis 75: Comparison: 7.5_(100)MF59 vs 15 Without MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio at day 202 = 2.388, 95% CI 2-sided [1.658 to 3.438]
Statistical Analysis 76: Comparison: 7.5_(100)MF59 vs 15_(50)MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio at day 202 = 0.987, 95% CI 2-sided [0.688 to 1.416]
Statistical Analysis 77: Comparison: 7.5_(100)MF59 vs 15_(100)MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio at day 202 = 1.012, 95% CI 2-sided [0.701 to 1.460]
Statistical Analysis 78: Comparison: 7.5_(100)MF59 vs 30 Without MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio at day 202 = 1.634, 95% CI 2-sided [1.128 to 2.366]
Statistical Analysis 79: Comparison: 15 Without MF59 vs 15_(50)MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio at day 202 = 0.413, 95% CI 2-sided [0.288 to 0.592]
Statistical Analysis 80: Comparison: 15 Without MF59 vs 15_(100)MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio at day 202 = 0.424, 95% CI 2-sided [0.294 to 0.610]
Statistical Analysis 81: Comparison: 15 Without MF59 vs 30 Without MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio at day 202 = 0.684, 95% CI 2-sided [0.473 to 0.990]
Statistical Analysis 82: Comparison: 15_(50)MF59 vs 15_(100)MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio at day 202 = 1.025, 95% CI 2-sided [0.714 to 1.473]
Statistical Analysis 83: Comparison: 15_(50)MF59 vs 30 Without MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio at day 202 = 1.656, 95% CI 2-sided [1.150 to 2.385]
Statistical Analysis 84: Comparison: 15_(100)MF59 vs 30 Without MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio at day 202 = 1.615, 95% CI 2-sided [1.115 to 2.339]
Statistical Analysis 85: Comparison: 3.75_(50)MF59 vs 7.5 Without MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio at day 387 = 1.906, 95% CI 2-sided [1.177 to 3.087]
Statistical Analysis 86: Comparison: 3.75_(50)MF59 vs 7.5_(50)MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio at day 387 = 0.945, 95% CI 2-sided [0.583 to 1.533]
Statistical Analysis 87: Comparison: 3.75_(50)MF59 vs 7.5_(100)MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio at day 387 = 0.763, 95% CI 2-sided [0.468 to 1.245]
Statistical Analysis 88: Comparison: 3.75_(50)MF59 vs 15 Without MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio at day 387 = 1.818, 95% CI 2-sided [1.119 to 2.956]
Statistical Analysis 89: Comparison: 3.75_(50)MF59 vs 15_(50)MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio at day 387 = 0.917, 95% CI 2-sided [0.568 to 1.481]
Statistical Analysis 90: Comparison: 3.75_(50)MF59 vs 15_(100)MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio at day 387 = 0.855, 95% CI 2-sided [0.524 to 1.396]
Statistical Analysis 91: Comparison: 3.75_(50)MF59 vs 30 Without MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio at day 387 = 1.203, 95% CI 2-sided [0.745 to 1.943]
Statistical Analysis 92: Comparison: 7.5 Without MF59 vs 7.5_(50)MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio at day 387 = 0.496, 95% CI 2-sided [0.310 to 0.794]
Statistical Analysis 93: Comparison: 7.5 Without MF59 vs 7.5_(100)MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio at day 387 = 0.400, 95% CI 2-sided [0.250 to 0.641]
Statistical Analysis 94: Comparison: 7.5 Without MF59 vs 15 Without MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio at day 387 = 0.954, 95% CI 2-sided [0.596 to 1.528]
Statistical Analysis 95: Comparison: 7.5 Without MF59 vs 15_(50)MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio at day 387 = 0.481, 95% CI 2-sided [0.306 to 0.758]
Statistical Analysis 96: Comparison: 7.5 Without MF59 vs 15_(100)MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio at day 387 = 0.449, 95% CI 2-sided [0.279 to 0.722]
Statistical Analysis 97: Comparison: 7.5 Without MF59 vs 30 Without MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio at day 387 = 0.631, 95% CI 2-sided [0.398 to 1.002]
Statistical Analysis 98: Comparison: 7.5_(50)MF59 vs 7.5_(100)MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio at day 387 = 0.807, 95% CI 2-sided [0.500 to 1.304]
Statistical Analysis 99: Comparison: 7.5_(50)MF59 vs 15 Without MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio at day 387 = 1.924, 95% CI 2-sided [1.193 to 3.102]
Statistical Analysis 100: Comparison: 7.5_(50)MF59 vs 15_(50)MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio at day 387 = 0.970, 95% CI 2-sided [0.611 to 1.541]
Statistical Analysis 101: Comparison: 7.5_(50)MF59 vs 15_(100)MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio at day 387 = 0.905, 95% CI 2-sided [0.561 to 1.460]
Statistical Analysis 102: Comparison: 7.5_(50)MF59 vs 30 Without MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio at day 387 = 1.273, 95% CI 2-sided [0.798 to 2.030]
Statistical Analysis 103: Comparison: 7.5_(100)MF59 vs 15 Without MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio at day 387 = 2.383, 95% CI 2-sided [1.474 to 3.851]
Statistical Analysis 104: Comparison: 7.5_(100)MF59 vs 15_(50)MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio at day 387 = 1.202, 95% CI 2-sided [0.754 to 1.915]
Statistical Analysis 105: Comparison: 7.5_(100)MF59 vs 15_(100)MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio at day 387 = 1.120, 95% CI 2-sided [0.689 to 1.821]
Statistical Analysis 106: Comparison: 7.5_(100)MF59 vs 30 Without MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio at day 387 = 1.576, 95% CI 2-sided [0.987 to 2.516]
Statistical Analysis 107: Comparison: 15 Without MF59 vs 15_(50)MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio at day 387 = 0.504, 95% CI 2-sided [0.316 to 0.805]
Statistical Analysis 108: Comparison: 15 Without MF59 vs 15_(100)MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio at day 387 = 0.470, 95% CI 2-sided [0.293 to 0.754]
Statistical Analysis 109: Comparison: 15 Without MF59 vs 30 Without MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio at day 387 = 0.662, 95% CI 2-sided [0.414 to 1.056]
Statistical Analysis 110: Comparison: 15_(50)MF59 vs 15_(100)MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio at day 387 = 0.932, 95% CI 2-sided [0.583 to 1.492]
Statistical Analysis 111: Comparison: 15_(50)MF59 vs 30 Without MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio at day 387 = 1.312, 95% CI 2-sided [0.831 to 2.071]
Statistical Analysis 112: Comparison: 15_(100)MF59 vs 30 Without MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric mean ratio at day 387 = 1.407, 95% CI 2-sided [0.880 to 2.249]
Statistical Analysis 113: Comparison: 3.75_(50)MF59 vs 7.5 Without MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric Mean Ratio at day 29 = 5.428, 95% CI 2-sided [4 to 7.365]
Statistical Analysis 114: Comparison: 3.75_(50)MF59 vs 7.5_(50)MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric Mean Ratio at day 29 = 1.091, 95% CI 2-sided [0.804 to 1.481]
Statistical Analysis 115: Comparison: 3.75_(50)MF59 vs 7.5_(100)MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric Mean Ratio at day 29 = 0.759, 95% CI 2-sided [0.559 to 1.031]
Statistical Analysis 116: Comparison: 3.75_(50)MF59 vs 15 Without MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric Mean Ratio at day 29 = 3.499, 95% CI 2-sided [2.577 to 4.751]
Statistical Analysis 117: Comparison: 3.75_(50)MF59 vs 15_(50)MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric Mean Ratio at day 29 = 0.982, 95% CI 2-sided [0.722 to 1.334]
Statistical Analysis 118: Comparison: 3.75_(50)MF59 vs 15_(100)MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric Mean Ratio at day 29 = 0.699, 95% CI 2-sided [0.513 to 0.95]
Statistical Analysis 119: Comparison: 3.75_(50)MF59 vs 30 Without MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric Mean Ratio at day 29 = 2.513, 95% CI 2-sided [1.846 to 3.421]
Statistical Analysis 120: Comparison: 7.5 Without MF59 vs 7.5_(50)MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric Mean Ratio at day 29 = 0.201, 95% CI 2-sided [0.149 to 0.272]
Statistical Analysis 121: Comparison: 7.5 Without MF59 vs 7.5_(100)MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric Mean Ratio at day 29 = 0.14, 95% CI 2-sided [0.103 to 0.189]
Statistical Analysis 122: Comparison: 7.5 Without MF59 vs 15 Without MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric Mean Ratio at day 29 = 0.645, 95% CI 2-sided [0.476 to 0.873]
Statistical Analysis 123: Comparison: 7.5 Without MF59 vs 15_(50)MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric Mean Ratio at day 29 = 0.181, 95% CI 2-sided [0.134 to 0.245]
Statistical Analysis 124: Comparison: 7.5 Without MF59 vs 15_(100)MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric Mean Ratio at day 29 = 0.129, 95% CI 2-sided [0.095 to 0.174]
Statistical Analysis 125: Comparison: 7.5 Without MF59 vs 30 Without MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric Mean Ratio at day 29 = 0.463, 95% CI 2-sided [0.341 to 0.628]
Statistical Analysis 126: Comparison: 7.5_(50)MF59 vs 7.5_(100)MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric Mean Ratio at day 29 = 0.696, 95% CI 2-sided [0.514 to 0.943]
Statistical Analysis 127: Comparison: 7.5_(50)MF59 vs 15 Without MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric Mean Ratio at day 29 = 3.207, 95% CI 2-sided [2.368 to 4.343]
Statistical Analysis 128: Comparison: 7.5_(50)MF59 vs 15_(50)MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric Mean Ratio at day 29 = 0.9, 95% CI 2-sided [0.665 to 1.218]
Statistical Analysis 129: Comparison: 7.5_(50)MF59 vs 15_(100)MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric Mean Ratio at day 29 = 0.64, 95% CI 2-sided [0.472 to 0.868]
Statistical Analysis 130: Comparison: 7.5_(50)MF59 vs 30 Without MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric Mean Ratio at day 29 = 2.303, 95% CI 2-sided [1.7 to 3.121]
Statistical Analysis 131: Comparison: 7.5_(100)MF59 vs 15 Without MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric Mean Ratio at day 29 = 4.608, 95% CI 2-sided [3.398 to 6.249]
Statistical Analysis 132: Comparison: 7.5_(100)MF59 vs 15_(50)MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric Mean Ratio at day 29 = 1.293, 95% CI 2-sided [0.954 to 1.753]
Statistical Analysis 133: Comparison: 7.5_(100)MF59 vs 15_(100)MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric Mean Ratio at day 29 = 0.92, 95% CI 2-sided [0.677 to 1.249]
Statistical Analysis 134: Comparison: 7.5_(100)MF59 vs 30 Without MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric Mean Ratio at day 29 = 3.31, 95% CI 2-sided [2.436 to 4.496]
Statistical Analysis 135: Comparison: 15 Without MF59 vs 15_(50)MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric Mean Ratio at day 29 = 0.281, 95% CI 2-sided [0.207 to 0.38]
Statistical Analysis 136: Comparison: 15 Without MF59 vs 15_(100)MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric Mean Ratio at day 29 = 0.2, 95% CI 2-sided [0.147 to 0.271]
Statistical Analysis 137: Comparison: 15 Without MF59 vs 30 Without MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric Mean Ratio at day 29 = 0.718, 95% CI 2-sided [0.529 to 0.975]
Statistical Analysis 138: Comparison: 15_(50)MF59 vs 15_(100)MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric Mean Ratio at day 29 = 0.712, 95% CI 2-sided [0.524 to 0.966]
Statistical Analysis 139: Comparison: 15_(50)MF59 vs 30 Without MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric Mean Ratio at day 29 = 2.56, 95% CI 2-sided [1.886 to 3.474]
Statistical Analysis 140: Comparison: 15_(100)MF59 vs 30 Without MF59; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric Mean Ratio at day 29 = 3.597, 95% CI 2-sided [2.646 to 4.89]

3. Secondary Outcome: Antibody Responses With and Without Seasonal Influenza Vaccination for Year 2009 to 2010.
Description: HI antibody assay (used to assess immune responses in subjects following vaccination) according to the Committee for Medicinal Products for Human Use (CHMP) guidance: in adults ages 18 to 60 years are:The percentage of subjects with seroconversion or significant increase in HI antibody is > 40%.The percentage of subjects achieving an HI titer ≥ 40 is > 70% and The GMR is > 2.5. All 3 criteria (seroconversion/significant increase, HI antibody titer ≥ 40, and GMR) had to be fulfilled to establish immunogenicity.Subgroup analysis based on receipt of recent seasonal vaccination. Comparison between subjects previously vaccinated versus not vaccinated with seasonal influenza vaccines.Subgroups without recent seasonal flu vaccine:PPS Day1, Day 1-22 and Day1-43 analysis set. N= 141, 147, 150, 148, 146, 146, 150, and 146 for Groups A, B, C, D, E, F, G, and H respectively. PPS Day 1-29 analysis set. N= 132, 140, 143, 139, 138, 136, 139, and 138 for Groups A, B, C, D, E, F, G,and H respectively.
Time Frame: Day 22, Day 29, Day 43
Population: The analysis was done on PPS population
Measure: Number (95% Confidence Interval); unit: percentage of Subjects
Arm/Group | 3.75_(50)MF59 | 7.5 Without MF59 | 7.5_(50)MF59 | 7.5_(100)MF59 | 15 Without MF59 | 15_(50)MF59 | 15_(100)MF59 | 30 Without MF59
Number analyzed (Participants) | 152 | 156 | 156 | 156 | 155 | 157 | 156 | 153
percentage of Subjects
  Seroconversion (Day 22/Day 1)with seasonal flu vac | 73 [39 to 94] | 22 [3 to 60] | 83 [36 to 100] | 100 [63 to 100] | 44 [14 to 79] | 73 [39 to 94] | 100 [54 to 100] | 71 [29 to 96]
  Seroconversion (Day 29/Day 1)with seasonal flu vac | 100 [72 to 100] | 67 [30 to 93] | 83 [36 to 100] | 100 [59 to 100] | 67 [30 to 93] | 100 [72 to 100] | 100 [48 to 100] | 83 [36 to 100]
  Seroconversion (Day 43/Day 1)with seasonal flu va | 91 [59 to 100] | 78 [40 to 97] | 67 [22 to 96] | 88 [47 to 100] | 78 [40 to 97] | 100 [72 to 100] | 100 [54 to 100] | 86 [42 to 100]
  HI titer ≥1:40 (Day 1)_ with seasonal flu vac | 18 [2 to 52] | 22 [3 to 60] | 50 [12 to 88] | 38 [9 to 76] | 0 [0 to 34] | 9 [0 to 41] | 17 [0 to 64] | 0 [0 to 41]
  HI titer ≥1:40 (Day 22)_ with seasonal flu vac | 73 [39 to 94] | 33 [7 to 70] | 100 [54 to 100] | 100 [63 to 100] | 44 [14 to 79] | 73 [39 to 94] | 100 [54 to 100] | 71 [29 to 96]
  HI titer ≥1:40 (Day 29)_ with seasonal flu vac | 100 [72 to 100] | 67 [30 to 93] | 100 [54 to 100] | 100 [59 to 100] | 67 [30 to 93] | 100 [72 to 100] | 100 [48 to 100] | 100 [54 to 100]
  HI titer ≥1:40 (Day 43)_ with seasonal flu vac | 100 [72 to 100] | 78 [40 to 97] | 100 [54 to 100] | 100 [63 to 100] | 78 [40 to 97] | 100 [72 to 100] | 100 [54 to 100] | 86 [42 to 100]
  Seroconversion (Day 22/Day 1)without flu vac | 82 [75 to 88] | 47 [39 to 55] | 77 [70 to 84] | 88 [81 to 93] | 59 [50 to 67] | 82 [75 to 88] | 91 [86 to 95] | 60 [51 to 68]
  Seroconversion (Day 29/Day 1)without flu vac | 98 [95 to 100] | 79 [71 to 85] | 99 [96 to 100] | 99 [95 to 100] | 88 [82 to 93] | 100 [97 to 100] | 100 [97 to 100] | 94 [89 to 97]
  Seroconversion (Day 43/Day 1)without flu vac | 99 [95 to 100] | 78 [70 to 84] | 98 [94 to 100] | 98 [94 to 100] | 85 [78 to 90] | 99 [95 to 100] | 99 [96 to 100] | 88 [82 to 93]
  HI titer ≥1:40 (Day 1) without flu vac | 10 [6 to 16] | 8 [4 to 14] | 11 [7 to 18] | 9 [5 to 15] | 16 [11 to 23] | 9 [5 to 15] | 7 [4 to 13] | 13 [8 to 20]
  HI titer ≥1:40 (Day 22)without flu vac | 84 [77 to 90] | 49 [41 to 57] | 80 [73 to 86] | 91 [85 to 95] | 62 [53 to 70] | 83 [76 to 89] | 93 [88 to 97] | 65 [57 to 73]
  HI titer ≥1:40 (Day 29) without flu vac | 99 [96 to 100] | 79 [72 to 86] | 100 [97 to 100] | 99 [95 to 100] | 90 [84 to 94] | 100 [97 to 100] | 100 [97 to 100] | 96 [92 to 99]
  HI titer ≥1:40 (Day 43) without flu vac | 99 [96 to 100] | 79 [71 to 85] | 100 [98 to 100] | 99 [95 to 100] | 88 [81 to 93] | 99 [96 to 100] | 100 [98 to 100] | 92 [86 to 96]

4. Secondary Outcome: Geometric Mean Titers (GMTs) With and Without Seasonal Influenza Vaccination for Year 2009 to 2010
Description: Immunogenicity was measured in terms of GMTs of Subgroups with receipt of recent seasonal vaccination. Comparison between subjects previously vaccinated versus not vaccinated with seasonal influenza vaccines
  Subgroups without recent seasonal flu vaccine:
  PPS Day 1, Day 1-22 and Day 1-43 analysis set. N= 141, 147, 150, 148, 146, 146, 150, and 146 for Groups A, B, C, D, E, F, G, and H respectively.
  PPS Day 1-29 analysis set. N= 132, 140, 143, 139, 138, 136, 139, and 138 for Groups A, B, C, D, E, F,G, and H respectively.
  Subgroups with recent seasonal flu vaccine:PPS Day 1-22 and Day 1-43 analysis set. N= 11, 9, 6, 8, 9, 11, 6, and 7 for Groups A, B, C, D, E, F, G,and H respectively.
  PPS Day 1-29 analysis set. N= 11, 9, 6, 7, 9, 11, 5, and 6 for Groups A, B, C, D, E, F, G, and H respectively
Time Frame: Day 1, Day 22, Day 29, Day 43
Population: The analysis was done on PPS population.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | 3.75_(50)MF59 | 7.5 Without MF59 | 7.5_(50)MF59 | 7.5_(100)MF59 | 15 Without MF59 | 15_(50)MF59 | 15_(100)MF59 | 30 Without MF59
Number analyzed (Participants) | 152 | 156 | 156 | 156 | 155 | 157 | 156 | 153
Titers
  Day 1_with seasonal flu vaccination | 6.22 [2.16 to 18] | 12 [3.63 to 42] | 22 [5.54 to 90] | 15 [4.5 to 47] | 5.42 [1.75 to 17] | 5.99 [2.16 to 17] | 15 [3.94 to 565] | 9.36 [2.69 to 33]
  Day 22_ with seasonal flu vaccination | 36 [9.11 to 146] | 44 [8.93 to 217] | 196 [32 to 1213] | 209 [45 to 976] | 48 [11 to 210] | 44 [11 to 166] | 345 [61 to 1961] | 111 [22 to 567]
  Day 29_ with seasonal flu vaccination | 278 [90 to 856] | 171 [47 to 625] | 785 [178 to 3450] | 1186 [317 to 4440] | 137 [41 to 457] | 670 [226 to 1988] | 771 [164 to 3628] | 184 [43 to 791]
  Day 43_ with seasonal flu vaccination | 260 [102 to 665] | 182 [62 to 537] | 503 [146 to 1729] | 594 [209 to 1687] | 81 [30 to 221] | 663 [268 to 1639] | 1035 [319 to 3363] | 228 [75 to 689]
  Day 1_without seasonal flu vaccination | 8.54 [7.03 to 10] | 7.08 [5.84 to 8.59] | 8.3 [6.86 to 10] | 7.76 [6.41 to 9.41] | 9.35 [7.71 to 11] | 7.47 [6.15 to 9.08] | 6.8 [5.61 to 8.24] | 9.1 [7.51 to 11]
  Day 22_ without seasonal flu vaccination | 115 [83 to 161] | 28 [20 to 38] | 85 [61 to 117] | 159 [115 to 220] | 52 [38 to 72] | 109 [79 to 152] | 158 [114 to 218] | 62 [45 to 85]
  Day 29_ without seasonal flu vaccination | 810 [633 to 1037] | 144 [113 to 183] | 669 [527 to 849] | 968 [760 to 1232] | 228 [179 to 291] | 756 [591 to 966] | 1080 [847 to 1377] | 297 [233 to 377]
  Day 43_ without seasonal flu vaccination | 600 [477 to 753] | 115 [92 to 144] | 477 [381 to 596] | 643 [514 to 805] | 182 [145 to 228] | 520 [414 to 653] | 770 [615 to 963] | 224 [179 to 281]

5. Secondary Outcome: Antibody Response Based on Baseline Seropositivity
Description: Subgroup analysis based on Subjects with seropositivity (pre-vaccination HI antibody titer < 1:10 and prevaccination HI antibody titer ≥ 1:10) at baseline.
  Subgroups with baseline HI titer < 1:10: PPS Day 1-29 analysis set. N= 104, 116, 111, 107, 109, 113,120, and 103 for Groups A, B, C, D, E, F, G, and H respectively.
  Subgroups with baseline HI titer ≥ 1:10: PPS Day 1-29 analysis set. N= 39, 33, 38, 39, 38, 34, 24, and 41 for Groups A, B, C, D, E, F, G, and H respectively.
Time Frame: Day 22, Day 29 and Day 43
Measure: Number (95% Confidence Interval); unit: percentage of Subjects
Arm/Group | 3.75_(50)MF59 | 7.5 Without MF59 | 7.5_(50)MF59 | 7.5_(100)MF59 | 15 Without MF59 | 15_(50)MF59 | 15_(100)MF59 | 30 Without MF59
Number analyzed (Participants) | 152 | 156 | 156 | 156 | 155 | 157 | 156 | 153
percentage of Subjects
  Seroconversion (Day 22/Day 1)_baseline HI < 1:10 | 81 [72 to 88] | 39 [30 to 48] | 79 [71 to 86] | 90 [84 to 95] | 54 [44 to 63] | 78 [69 to 85] | 92 [86 to 96] | 61 [52 to 70]
  Seroconversion (Day 29/Day 1)_baseline HI < 1:10 | 99 [95 to 100] | 75 [66 to 83] | 100 [97 to 100] | 98 [93 to 100] | 85 [77 to 91] | 100 [97 to 100] | 100 [97 to 100] | 97 [92 to 99]
  Seroconversion (Day 43/Day 1)_baseline HI < 1:10 | 99 [95 to 100] | 75 [67 to 83] | 100 [97 to 100] | 98 [94 to 100] | 83 [75 to 90] | 99 [95 to 100] | 100 [97 to 100] | 91 [84 to 96]
  HI titer ≥1:40 (Day 1)_ baseline HI <1:10 | 0 [0 to 3] | 0 [0 to 3] | 0 [0 to 3] | 0 [0 to 3] | 0 [0 to 3] | 0 [0 to 3] | 0 [0 to 3] | 0 [0 to 3]
  HI titer ≥1:40 (Day 22)_ baseline HI <1:10 | 81 [72 to 88] | 39 [30 to 48] | 79 [71 to 86] | 90 [84 to 95] | 54 [44 to 63] | 78 [69 to 85] | 92 [86 to 96] | 61 [52 to 70]
  HI titer ≥1:40 (Day 29)_ baseline HI <1:10 | 99 [95 to 100] | 75 [66 to 83] | 100 [97 to 100] | 98 [93 to 100] | 85 [77 to 91] | 100 [97 to 100] | 100 [97 to 100] | 97 [92 to 99]
  HI titer ≥1:40 (Day 43)_ baseline HI <1:10 | 99 [95 to 100] | 75 [67 to 83] | 100 [97 to 100] | 98 [94 to 100] | 83 [75 to 90] | 99 [95 to 100] | 100 [97 to 100] | 91 [84 to 96]
  Seroconversion (Day 22/Day 1)_baseline HI ≥ 1:10 | 83 [69 to 93] | 69 [51 to 83] | 73 [57 to 86] | 83 [68 to 93] | 71 [54 to 84] | 95 [82 to 99] | 89 [72 to 98] | 57 [41 to 72]
  Seroconversion (Day 29/Day 1)_baseline HI ≥ 1:10 | 97 [87 to 100] | 88 [72 to 97] | 95 [82 to 99] | 100 [91 to 100] | 92 [79 to 98] | 100 [90 to 100] | 100 [86 to 100] | 85 [71 to 94]
  Seroconversion (Day 43/Day 1)_baseline HI ≥ 1:10 | 95 [84 to 99] | 86 [70 to 95] | 88 [74 to 96] | 95 [83 to 99] | 88 [74 to 96] | 97 [86 to 100] | 96 [82 to 100] | 81 [66 to 91]
  HI titer ≥1:40 (Day 1)_ baseline HI ≥1:10 | 38 [24 to 54] | 40 [24 to 58] | 49 [33 to 65] | 41 [26 to 58] | 59 [42 to 74] | 38 [22 to 55] | 43 [24 to 63] | 45 [30 to 61]
  HI titer ≥1:40 (Day 22)_ baseline HI ≥1:10 | 90 [77 to 97] | 80 [63 to 92] | 85 [71 to 94] | 93 [80 to 98] | 80 [65 to 91] | 97 [86 to 100] | 100 [88 to 100] | 76 [61 to 88]
  HI titer ≥1:40 (Day 29)_ baseline HI ≥1:10 | 100 [91 to 100] | 91 [76 to 98] | 100 [91 to 100] | 100 [91 to 100] | 97 [86 to 100] | 100 [90 to 100] | 100 [86 to 100] | 95 [83 to 99]
  HI titer ≥1:40 (Day 43)_ baseline HI ≥1:10 | 100 [92 to 100] | 91 [77 to 98] | 100 [91 to 100] | 100 [91 to 100] | 98 [87 to 100] | 100 [91 to 100] | 100 [88 to 100] | 93 [81 to 99]

6. Secondary Outcome: Geometric Mean Titers (GMTs) Based on Baseline Seropositivity
Description: Subgroup analysis based on Subjects with seropositivity (pre-vaccination HI antibody titer < 1:10 and prevaccination HI antibody titer ≥ 1:10) at baseline.
  Immunogenicity responses in subjects who are seropositive (A/H1N1 2009 HI titer ≥ 1:10) at Baseline [Day 1 (pre-vaccination)] as compared to those who are seronegative (HI titer < 1:10).
Time Frame: Day 1, Day 22, Day 29, Day 43
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | 3.75_(50)MF59 | 7.5 Without MF59 | 7.5_(50)MF59 | 7.5_(100)MF59 | 15 Without MF59 | 15_(50)MF59 | 15_(100)MF59 | 30 Without MF59
Number analyzed (Participants) | 152 | 156 | 156 | 156 | 155 | 157 | 156 | 153
Titers
  GMTDay 1 HI <1:10(110,121,115,115,114,120,128,11 | 5 [5 to 5.1] | 5 [5 to 5.1] | 5.1 [5 to 5.1] | 5.1 [5 to 5.1] | 5 [5 to 5.1] | 5 [5 to 5.07] | 5.1 [5 to 5.2] | 5.1 [5 to 5.2]
  GMTDay 22 HI<1:10(110,121,115,115,114,120,128,11 | 80 [57 to 111] | 18 [13 to 25] | 62 [45 to 85] | 130 [94 to 180] | 26 [19 to 36] | 72 [52 to 98] | 130 [96 to 177] | 39 [28 to 54]
  GMTDay 29HI <1:10(110,121,115,115,114,120,128,11 | 664 [505 to 872] | 100 [78 to 130] | 638 [490 to 830] | 885 [676 to 1157] | 149 [114 to 194] | 685 [527 to 890] | 950 [736 to 1227] | 234 [179 to 307]
  GMTDay 43HI <1:10(110,121,115,115,114,120,128,11 | 490 [381 to 630] | 85 [67 to 108] | 437 [342 to 559] | 568 [444 to 727] | 121 [95 to 155] | 463 [363 to 590] | 717 [566 to 908] | 177 [138 to 227]
  GMT Day 1 HI ≥ 1:10(42,35,41,41,41,37,28,42) | 40 [28 to 57] | 32 [21 to 47] | 47 [32 to 68] | 32 [22 to 46] | 52 [36 to 75] | 35 [24 to 52] | 40 [26 to 63] | 48 [33 to 69]
  GMT Day 22_HI ≥1:10(42,35,41,41,41,37,28,42) | 343 [187 to 628] | 132 [68 to 258] | 311 [164 to 590] | 320 [171 to 599] | 284 [151 to 532] | 417 [217 to 802] | 460 [219 to 965] | 252 [134 to 475]
  GMT Day 29_HI ≥1:10(42,35,41,41,41,37,28,42) | 1178 [782 to 1776] | 460 [294 to 721] | 1063 [689 to 1640] | 1281 [843 to 1948] | 543 [356 to 830] | 1197 [771 to 1857] | 2088 [1240 to 3516] | 641 [422 to 973]
  GMT Day 43_HI ≥1:10(42,35,41,41,41,37,28,42) | 876 [604 to 1271] | 320 [212 to 482] | 657 [443 to 974] | 881 [599 to 1295] | 464 [316 to 684] | 838 [561 to 1253] | 1184 [751 to 1867] | 428 [290 to 631]

7. Secondary Outcome: Number of Subjects Reporting Solicited Local and Systemic Symptoms After the First Vaccination
Description: Solicited local and systemic reactions were assessed after the first vaccination by vaccine group. Source Vocabulary Name: MedDRA (13.1).
Time Frame: 7 days after first vaccination
Population: The analysis was performed on safety set population
Measure: Number; unit: Participants
Arm/Group | 3.75_(50)MF59 | 7.5 Without MF59 | 7.5_(50)MF59 | 7.5_(100)MF59 | 15 Without MF59 | 15_(50)MF59 | 15_(100)MF59 | 30 Without MF59
Number analyzed (Participants) | 171 | 167 | 167 | 168 | 167 | 168 | 166 | 165
Participants
  Pain | 62 | 43 | 52 | 86 | 47 | 65 | 72 | 51
  Erythema | 3 | 2 | 4 | 3 | 1 | 1 | 6 | 5
  Swelling | 8 | 5 | 5 | 7 | 11 | 11 | 10 | 6
  Induration | 14 | 5 | 10 | 12 | 10 | 11 | 15 | 12
  Tenderness | 72 | 49 | 59 | 96 | 50 | 78 | 69 | 60
  Chills | 8 | 3 | 9 | 11 | 5 | 8 | 8 | 8
  Myalgia | 16 | 8 | 13 | 27 | 8 | 15 | 17 | 12
  Arthralgia | 7 | 3 | 9 | 7 | 3 | 8 | 7 | 3
  Headache | 24 | 15 | 30 | 37 | 16 | 25 | 27 | 17
  Nausea | 10 | 14 | 13 | 14 | 7 | 11 | 12 | 9
  Vomiting | 4 | 5 | 10 | 4 | 5 | 8 | 5 | 5
  Diarrhoea | 12 | 7 | 6 | 2 | 10 | 3 | 4 | 6
  Fatigue | 27 | 17 | 23 | 29 | 17 | 23 | 29 | 16
  Fever | 9 | 10 | 13 | 14 | 9 | 17 | 16 | 7
  Stayed home | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0
  Analgesic./anti pyretic used | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: Number of Subjects Reporting Solicited Local and Systemic Symptoms After the Second Vaccination
Description: Solicited local and systemic reactions were assessed after the second vaccination by vaccine group.Source Vocabulary Name: MedDRA (13.1)
Time Frame: 7 days after second vaccination
Population: The analysis was performed on safety set population
Measure: Number; unit: Participant
Arm/Group | 3.75_(50)MF59 | 7.5 Without MF59 | 7.5_(50)MF59 | 7.5_(100)MF59 | 15 Without MF59 | 15_(50)MF59 | 15_(100)MF59 | 30 Without MF59
Number analyzed (Participants) | 165 | 163 | 164 | 163 | 162 | 167 | 162 | 164
Participant
  Pain | 53 | 35 | 46 | 59 | 42 | 57 | 48 | 50
  Erythema | 4 | 1 | 4 | 5 | 5 | 4 | 5 | 5
  Swelling | 8 | 5 | 10 | 9 | 11 | 10 | 12 | 10
  Induration | 10 | 2 | 9 | 6 | 9 | 15 | 13 | 10
  Tenderness | 55 | 42 | 50 | 65 | 38 | 67 | 57 | 54
  Chills | 7 | 5 | 5 | 4 | 7 | 4 | 3 | 3
  Myalgia | 12 | 4 | 9 | 16 | 6 | 8 | 9 | 15
  Arthralgia | 2 | 0 | 1 | 4 | 2 | 2 | 0 | 2
  Headache | 12 | 12 | 12 | 19 | 14 | 11 | 13 | 9
  Nausea | 11 | 7 | 5 | 6 | 8 | 16 | 4 | 5
  Vomiting | 6 | 3 | 4 | 7 | 3 | 3 | 3 | 3
  Diarrhoea | 6 | 6 | 5 | 5 | 7 | 7 | 2 | 4
  Fatigue | 16 | 11 | 15 | 14 | 17 | 10 | 13 | 6
  Fever | 10 | 6 | 5 | 5 | 10 | 8 | 7 | 4
  Stayed home | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Analgesic/anti pyretic used | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

9. Secondary Outcome: Number of Participants Reporting Unsolicited Adverse Events (AEs)
Description: Safety was measured in terms of the Number of Participants Reporting Unsolicited AEs. Source Vocabulary Name: MedDRA (13.1)
Time Frame: Safety monitoring periods were the Primary Period: Day 1 (1st vaccination) through ≤21 days post second vaccination, and the Follow-up Period: >21 Days post second vaccination to 12 months after second vaccination
Population: The analysis was done on unsolicited safety set population.
Measure: Number; unit: Subjects
Arm/Group | 3.75_(50)MF59 | 7.5 Without MF59 | 7.5_(50)MF59 | 7.5_(100)MF59 | 15 Without MF59 | 15_(50)MF59 | 15_(100)MF59 | 30 Without MF59
Number analyzed (Participants) | 171 | 168 | 169 | 168 | 168 | 168 | 167 | 169
Subjects
  AEs: all (Days 1-43) | 98 | 80 | 80 | 85 | 86 | 93 | 79 | 79
  SAEs: all (Days 1-43) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  AEs leading to premature withdrawal (Days 1-43) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  AEs leading to new onset of chronic disorder | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  AE leading to medically attended visits(Days 1-43) | 31 | 34 | 25 | 40 | 34 | 35 | 28 | 24
  AEs: all (Days 44-387) | 95 | 98 | 102 | 93 | 90 | 101 | 90 | 95
  SAEs: all (Days 44-387) | 0 | 5 | 6 | 4 | 3 | 4 | 1 | 0
  AEs leading to premature withdrawal (Days 44-387) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  AEs leading to new onset of chronic dis. | 2 | 7 | 4 | 3 | 4 | 3 | 6 | 3
  AE leading to medically attended visit(Days44-387) | 95 | 97 | 102 | 93 | 90 | 100 | 89 | 95

ADVERSE EVENTS:
Time Frame: All adverse events (AEs) and serious adverse events (SAEs) were collected for the whole study (study day 1 to day 387).
Description: If the adverse event was solicited then the assessment was entered as systematic. However, if the adverse event was not solicited (unsolicited), then the assessment was entered as non-systematic.
Arm/Group | 3.75_(50)MF59 | 7.5 Without MF59 | 7.5_(50)MF59 | 7.5_(100)MF59 | 15 Without MF59 | 15_(50)MF59 | 15_(100)MF59 | 30 Without MF59
Serious Adverse Events (participants affected / at risk) | 0/171 | 5/168 | 7/169 | 4/168 | 3/168 | 4/168 | 1/167 | 0/169
Other Adverse Events (participants affected / at risk) | 171/171 | 168/168 | 169/169 | 168/168 | 168/168 | 168/168 | 167/167 | 169/169
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 3.75_(50)MF59 (N=171) | 7.5 Without MF59 (N=168) | 7.5_(50)MF59 (N=169) | 7.5_(100)MF59 (N=168) | 15 Without MF59 (N=168) | 15_(50)MF59 (N=168) | 15_(100)MF59 (N=167) | 30 Without MF59 (N=169)
Febrile Convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hydrocele (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cerumen Impaction (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Appendicitis Perforated (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chronic Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Otitis Media Chronic (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Peritonsillar Abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pharyngitis Streptococcal (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pharyngotonsillitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Staphylococcal Scalded Skin Syndrome (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Viral Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Altered state of consciousness (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Foreign Body (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ulna Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Aggression (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bipolar Disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Intermittent Explosive Disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oppositional Defiant Disorder (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Post-Traumatic Stress Disorder (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ovarian Mass (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pharyngeal Stenosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Swelling Face (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 3.75_(50)MF59 (N=171) | 7.5 Without MF59 (N=168) | 7.5_(50)MF59 (N=169) | 7.5_(100)MF59 (N=168) | 15 Without MF59 (N=168) | 15_(50)MF59 (N=168) | 15_(100)MF59 (N=167) | 30 Without MF59 (N=169)
Cough (Respiratory, thoracic and mediastinal disorders) | 34 | 36 | 30 | 27 | 34 | 35 | 40 | 38
Nasopharyngitis (Infections and infestations) | 14 | 4 | 10 | 10 | 7 | 10 | 9 | 7
Pyrexia (General disorders) | 41 | 34 | 38 | 34 | 44 | 34 | 34 | 26
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 10 | 9 | 7 | 9 | 11 | 17 | 15 | 11
Upper respiratory track infection (Infections and infestations) | 29 | 36 | 23 | 26 | 25 | 21 | 21 | 22
Vomiting (Gastrointestinal disorders) | 22 | 14 | 27 | 20 | 19 | 18 | 20 | 21
Injection site pain (General disorders) | 98 | 70 | 85 | 117 | 85 | 99 | 100 | 89
Headache (Nervous system disorders) | 37 | 31 | 39 | 44 | 28 | 37 | 38 | 28
Injection site erythema (General disorders) | 29 | 16 | 26 | 38 | 25 | 26 | 36 | 35
Myalgia (Musculoskeletal and connective tissue disorders) | 24 | 10 | 17 | 36 | 13 | 18 | 22 | 22
Fatigue (General disorders) | 33 | 22 | 31 | 32 | 30 | 29 | 36 | 20
Injection site induration (General disorders) | 23 | 5 | 19 | 19 | 18 | 23 | 32 | 24
Nausea (Gastrointestinal disorders) | 21 | 20 | 13 | 19 | 16 | 23 | 16 | 14
Diarrhea (Gastrointestinal disorders) | 22 | 16 | 17 | 10 | 22 | 13 | 12 | 16
Injection site swelling (General disorders) | 17 | 8 | 14 | 19 | 19 | 20 | 24 | 18
Chills (General disorders) | 17 | 8 | 13 | 14 | 12 | 12 | 11 | 11
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 2 | 12 | 9 | 6 | 9 | 8 | 4
Conjunctivitis (Infections and infestations) | 3 | 5 | 4 | 15 | 6 | 7 | 5 | 5
Bronchitis (Infections and infestations) | 13 | 8 | 5 | 10 | 7 | 4 | 6 | 3
Pharyngitis (Infections and infestations) | 13 | 9 | 14 | 15 | 12 | 10 | 6 | 6
Pharyngitis Streptococcal (Infections and infestations) | 17 | 19 | 18 | 20 | 15 | 20 | 13 | 17
Sinusitis (Infections and infestations) | 9 | 7 | 7 | 11 | 9 | 13 | 3 | 9
Viral Infection (Infections and infestations) | 13 | 5 | 11 | 13 | 10 | 17 | 13 | 12
Asthma (Respiratory, thoracic and mediastinal disorders) | 14 | 8 | 10 | 10 | 6 | 7 | 11 | 6
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 12 | 7 | 6 | 4 | 11 | 6 | 8 | 8
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 13 | 9 | 5 | 11 | 12 | 12 | 14 | 5
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 10 | 9 | 7 | 9 | 11 | 17 | 15 | 11
Otitis Media (Infections and infestations) | 17 | 14 | 28 | 18 | 21 | 18 | 23 | 23
OTITIS MEDIA ACUTE (Infections and infestations) | 9 | 3 | 4 | 4 | 7 | 3 | 5 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No